CLINICAL TRIAL: NCT00900029
Title: A Twenty-Four Week Non-Interventional Safety Follow-Up to HP 802-247-09-015
Brief Title: Safety Follow-Up to HP 802-247-09-015
Status: Completed | Type: Observational
Sponsor: Healthpoint (Industry)
Responsible Party: Sponsor
Other Study IDs: 802-247-09-016
Record Dates: First submitted 2009-05-11; First posted 2009-05-12 (Estimated); Results first posted 2016-09-29 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2016-09

CONDITIONS: Venous Leg Ulcer; Venous Stasis Ulcer
Keywords: Venous Leg Ulcer; Venous Stasis Ulcer; VLU; VSU; Leg Ulcer; Leg Wound
MeSH Terms: conditions — Varicose Ulcer; Leg Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- No HP802 Treatment: Treatment received in Study 802-247-09-015 was HP802
  Interventions: Biological: No HP802 Treatment
- No HP802 Vehicle Treatment: Treatment received in Study 802-247-09-015 was HP802 Vehicle
  Interventions: Other: No HP802 Vehicle Treatment

INTERVENTIONS:
Biological: No HP802 Treatment
  Groups: No HP802 Treatment
Other: No HP802 Vehicle Treatment
  Groups: No HP802 Vehicle Treatment

SUMMARY:
This is a 24-week observational follow safety study for Study 802-247-09-015.

DETAILED DESCRIPTION:
The objective of this study is to examine the durability of previous target wound closures, identify new test article-related adverse events, record new target wound closures, and examine ongoing adverse events not resolved in subjects who participated in HP 802-247-09-015.

ELIGIBILITY:
INCLUSION CRITERIA:

* Provide informed consent
* Willing to comply with protocol instructions, including allowing all study assessments.
* Subject was randomized in HP 802-247-09-015 and received at least one application of a test article, whether active or placebo.
* Subject has ended their participation in HP 802-247-09-015 by virtue of completing the study, or by dropping out prior to completion.

Exclusion Criteria

* Subjects who refuse to provide written informed consent will be excluded from this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who participated in Study No. 802-247-09-015 - "A Phase II Randomized, Double Blind, Placebo Controlled Dose Finding Study Investigating the Efficacy of HP802-247 in Venous Leg Ulcers" and agreed to continue with the follow-up study.
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2009-06; Primary Completion 2011-10 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hebert B Slade, MD, FAAAAI, Study Director — Healthpoint
Locations (30):
- United States (29):
  - University of AZ College of Medicine, Tucson, Arizona
  - Center for Clinical Research, Castro Valley, California
  - ILD Consulting, Inc., Encinitas, California
  - Vascular Surgery Associates, Los Angeles, California
  - UCSD Wound Treatment and Research Center, San Diego, California
  - University of Miami, Miami, Florida
  - Doctors Research Network, South Miami, Florida
  - Robert J. Snyder, Tamarac, Florida
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Passavant Area Hospital, Jacksonville, Illinois
  - Rosalind Franklin University, North Chicago, Illinois
  - Southern Illinois University, Springfield, Illinois
  - Johns Hopkins Wound Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - New England Sinai Hospital, Stoughton, Massachusetts
  - Advanced Foot and Ankle Center, Las Vegas, Nevada
  - Vincent Giacalone, Emerson, New Jersey
  - St. Luke's Roosevelt Hospital Center, New York, New Jersey
  - Overglook Hospital Wound Healing Program, Summit, New Jersey
  - University of North Carolina, Chapel Hill, North Carolina
  - Harrisburg Foot and Ankle Center, Harrisburg, Pennsylvania
  - Center for Advanced Wound Care, Reading, Pennsylvania
  - Arlington Research Center, Arlington, Texas
  - Wound Care Consultants, Dallas, Texas
  - Southwest Regional Wound Care Center, Lubbock, Texas
  - Peripheral Vascular Associates, San Antonio, Texas
  - Dixie Regional Medical Center's Wound Clinic, St. George, Utah
  - Lake Washington Vascular, PLLC, Bellevue, Washington
  - Providence Sacred Heart Medical Center Wound Clinic, Spokane, Washington
- Aging Rehabilitation & Geriatric Care Research Center, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible subjects were those who completed study 802-247-09-015. Of the 228 subjects who completed 802-247-09-015, 206 consented to enter this safety follow up study, between June 1, 2009 and October, 20, 2011.
Pre-assignment Details: Both PIs and subjects remained blinded to the therapy each subject received in 802-247-09-015. No test article was administered during this study and any therapy was at the discretion of the PI, with no restrictions.
Groups:
- LD-Q14D: LD-Q14D: 0.5 x 106 cell/mL applied to wound surface every 2 weeks
- LD-Q7D: LD-Q7D: 0.5 x 106 cell/mL applied to wound surface every week
- HD-Q14D: HD-Q14D: 5.0 x 106 cell/mL applied to wound surface every 2 weeks
- HD-Q7D: HD-Q7D: 5.0 x 106 cell/mL applied to wound surface every week
- HP802-247 Vehicle: Acellular vehicle applied weekly applied to wound surface every week
Period: Overall Study
Arm/Group | LD-Q14D | LD-Q7D | HD-Q14D | HD-Q7D | HP802-247 Vehicle
Started | 38 | 41 | 41 | 42 | 44
Completed | 35 | 37 | 38 | 35 | 38
Not Completed | 3 | 4 | 3 | 7 | 6
Not completed — Lost to Follow-up | 0 | 2 | 1 | 4 | 4
Not completed — Withdrawal by Subject | 2 | 2 | 1 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 1
Not completed — Death | 1 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Subjects and PIs remained blinded as treatment in the 802-247-09-015 study. There were no restrictions as to treatment by the PIs during this study. Blinding was maintained in order to assess the final outcomes of this study in relation to the therapy received in the prior study
Groups:
- HP802-247 Vehicle: Acellular vehicle applied weekly
- Total: Total of all reporting groups
Arm/Group | HP802-247 Vehicle | LD-Q14D | LD-Q7D | HD-Q14D | HD-Q7D | Total
Number analyzed (Participants) | 44 | 38 | 41 | 41 | 42 | 206
Age, Customized [Number; unit: participants]
  18-39 years | 1 | 4 | 3 | 3 | 4 | 15
  40-49 years | 8 | 6 | 4 | 6 | 6 | 30
  50-59 years | 11 | 7 | 10 | 8 | 6 | 42
  60+ years | 24 | 21 | 24 | 24 | 26 | 119
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 13 | 19 | 20 | 84
  Male | 29 | 21 | 28 | 22 | 22 | 122
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 11 | 10 | 6 | 12 | 48
  Not Hispanic or Latino | 35 | 27 | 31 | 35 | 30 | 158
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 9 | 8 | 9 | 11 | 8 | 45
  White | 31 | 29 | 28 | 29 | 30 | 147
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4 | 1 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Closed Target Ulcers at Each Visit
Description: At each visit the status of closed target ulcers was evaluated as remained closed or re-opened.
Time Frame: Over the 24-week study period, at each of the bi-monthly visits
Population: Subjects who completed the 802-247-09-015 study with a closed target wound attended three bimonthly visits.
Measure: Number; unit: participants
Arm/Group | LD-Q14D | LD-Q7D | HD-Q14D | HD-Q7D | HP802-247 Vehicle
Number analyzed (Participants) | 27 | 21 | 25 | 23 | 18
participants
  Enrollment | 27 | 21 | 25 | 23 | 18
  Month 2 (Visit 1) | 22 | 19 | 24 | 20 | 17
  Month 4 (Visit 2) | 25 | 19 | 22 | 21 | 16
  Month 6 (Visit 3) | 25 | 19 | 21 | 20 | 15

2. Primary Outcome: Number of Subjects With Target Wound Closed for the First Time During the Study Period.
Description: At each visit the status of open target ulcers was evaluated as "remained open" or "closed".
Time Frame: Over the 24-week study period, at each of the bi-monthly visits
Population: Subjects who completed the 802-247-09-015 study with open target wound attended three bimonthly visits over the duration of the study.
Measure: Number; unit: participants
Arm/Group | LD-Q14D | LD-Q7D | HD-Q14D | HD-Q7D | HP802-247 Vehicle
Number analyzed (Participants) | 8 | 16 | 13 | 12 | 20
participants
  Month 2 (Visit 1) | 3 | 1 | 4 | 2 | 4
  Month 4 (Visit 2) | 5 | 3 | 4 | 5 | 8
  Month 6 (Visit 3) | 4 | 4 | 7 | 6 | 7

ADVERSE EVENTS:
Time Frame: The duration of the 24-week study period
Description: All subjects with at least one study visit were questioned about adverse events and were included in the number of participants assessed for safety. The first assessments at each visit were about changes in general health and concomitant medications and the occurrence of adverse events.
Arm/Group | LD-Q14D | LD-Q7D | HD-Q14D | HD-Q7D | HP802-247 Vehicle
Serious Adverse Events (participants affected / at risk) | 3/38 | 0/41 | 4/41 | 5/42 | 4/44
Other Adverse Events (participants affected / at risk) | 10/38 | 6/41 | 5/41 | 11/42 | 14/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LD-Q14D (N=38) | LD-Q7D (N=41) | HD-Q14D (N=41) | HD-Q7D (N=42) | HP802-247 Vehicle (N=44)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alcohol detoxification (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aneurysm ruptured (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous insufficiency (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LD-Q14D (N=38) | LD-Q7D (N=41) | HD-Q14D (N=41) | HD-Q7D (N=42) | HP802-247 Vehicle (N=44)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Wound infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (2) | 2 (3) | 2 (4)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 4 (5) | 2 (2) | 0 (0) | 3 (4) | 6 (9)
Infections and infestations (Infections and infestations) | 5 (6) | 2 (2) | 1 (2) | 5 (7) | 7 (10)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 4 (6) | 3 (3) | 2 (4) | 4 (5) | 9 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less